CLINICAL TRIAL: NCT03012880
Title: Phase 2 Trial of Ixazomib, Lenalidomide, Dexamethasone, and Daratumumab in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Ixazomib Citrate, Lenalidomide, Dexamethasone, and Daratumumab in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1686; NCI-2017-00007 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1686 (Other: Mayo Clinic); 16-006835 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-06

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib, lenalidomide, daratumumab, dexamethasone) (Experimental): INDUCTION PHASE: Patients receive ixazomib citrate PO on days 1, 8, and 15 and lenalidomide PO on days 1-21. Patients receive daratumumab IV over 3-7 hours on days 1, 8, 15, and 22 of courses 1 and 2, on days 1 and 15 of courses 3, 4, and 5, and on day 1 of courses 7 and beyond. Patients also receive dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive ixazomib citrate PO on days 1, 8, and 15 and daratumumab IV over 3-7 hours on day 1. Courses repeat every 28 days for up to 36 months from registration in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well ixazomib citrate, lenalidomide, dexamethasone, and daratumumab work in treating patients with newly diagnosed multiple myeloma. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as lenalidomide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as daratumumab, may block cancer growth in different ways by targeting certain cells. Giving ixazomib citrate, lenalidomide, dexamethasone, and daratumumab may work better in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate (CR) of the four-drug combination of ixazomib, lenalidomide, dexamethasone and daratumumab in patients with previously untreated symptomatic multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR), and very good partial response (VGPR) rate with the four drug combination of ixazomib, lenalidomide, dexamethasone and daratumumab, when used as initial therapy in patients with previously untreated symptomatic MM.

II. To determine the progression free survival and overall survival among patients with previously untreated symptomatic MM following treatment with the four drug combination of Ixazomib, lenalidomide, dexamethasone and daratumumab followed by ixazomib and daratumumab maintenance till progression.

II. To determine the toxicities associated with the four drug combination of ixazomib, lenalidomide, dexamethasone and daratumumab in patients with previously untreated symptomatic MM.

TERTIARY OBJECTIVES:

I. To examine the proportion of minimal residual disease (MRD) negativity following induction therapy with the four-drug combination of ixazomib, lenalidomide, dexamethasone and daratumumab.

II. To assess the quality of life using patient completed Functional Assessment of Cancer Treatment (FACT)/Gynecologic Oncology Group (GOG) questionnaires.

OUTLINE:

INDUCTION PHASE: Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15 and lenalidomide PO on days 1-21. Patients receive daratumumab intravenously (IV) over 3-7 hours on days 1, 8, 15, and 22 of courses 1 and 2, on days 1 and 15 of courses 3, 4, and 5, and on day 1 of courses 7 and beyond. Patients also receive dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive ixazomib citrate PO on days 1, 8, and 15 and daratumumab IV over 3-7 hours on day 1. Courses repeat every 28 days for up to 36 months from registration in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 or 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Untransfused platelet count >= 75000/mm^3
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Previously untreated for myeloma or have received no more than one cycle of any treatment regimen; NOTE: Prior radiation therapy for the treatment of solitary plasmacytoma is permitted; prior therapy with clarithromycin, dehydroepiandrosterone (DHEA), anakinra, pamidronate or zoledronic acid is permitted; any additional agents not listed must be approved by the principal investigator
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures

  * Female patients: if they are of childbearing potential, agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to follow the requirements of the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Willing to provide bone marrow and blood samples for planned research

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma
* Diagnosed or treated for another malignancy =< 2 years prior to registration or previously diagnosed with another malignancy and have any evidence of residual disease; NOTE: Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, or any ancillary therapy considered investigational; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Peripheral neuropathy >= grade 2 on clinical examination or grade 1 with pain during the screening period
* Major surgery =< 14 days prior to registration
* Systemic treatment with strong CYP3A4 inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, St. John's wort) =< 14 days prior to registration
* Evidence of current uncontrolled cardiovascular conditions, including hypertension, cardiac arrhythmias, congestive heart failure, unstable angina, or myocardial infarction =< 6 months; Note: Prior to entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant
* Radiotherapy =< 14 days prior to registration; NOTE: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or investigator's brochure), or known sensitivity to mammalian-derived products
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib, lenalidomide or dexamethasone including difficulty swallowing
* Diarrhea > grade 1, based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grading, in the absence of antidiarrheals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A; Cohort B: INDUCTION PHASE: Patients receive ixazomib citrate PO on days 1, 8, and 15 and lenalidomide PO on days 1-21. Patients receive daratumumab IV over 3-7 hours on days 1, 8, 15, and 22 of courses 1 and 2, on days 1 and 15 of courses 3, 4, and 5, and on day 1 of courses 7 and beyond. Patients also receive dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.>
  > MAINTENANCE PHASE: Patients receive ixazomib citrate PO on days 1, 8, and 15 and daratumumab IV over 3-7 hours on day 1. Courses repeat every 28 days for up to 36 months from registration in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 40 | 40
Completed | 38 | 40
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 81] | 64.5 [33 to 81] | 63.5 [33 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 18 | 25 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 36 | 72
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 37 | 38 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve a Confirmed Complete Response (CR)
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 40
proportion of participants | 0.32 [0.184 to 0.474] | 0.30 [0.175 to 0.475]

2. Secondary Outcome: Proportion of Patients That Experienced a Grade 3 or Higher Adverse Event.
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables are in the adverse event section of this report. The rate of patients that suffered a grade 3 or higher adverse event are reported here.
Time Frame: 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 40
proportion of participants | 0.58 | 0.53

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Will be estimated by the number of patients who achieve a stringent complete response (sCR), CR, VGPR or partial response (PR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportions will be calculated.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 40
proportion of participants | 0.97 [0.87 to 1.00] | 0.95 [0.83 to 1.00]

4. Secondary Outcome: Overall Survival (OS)
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 40
Months | NA [NA to NA] — Too few events observed, can't calculate median or limits. | NA [NA to NA] — Too few events observed, can't calculate median or limits.

5. Secondary Outcome: Progression Free Survival
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 40
Months | NA [NA to NA] — Too few events observed, can't calculate median or limits. | NA [NA to NA] — Too few events observed, can't calculate median or limits.

6. Secondary Outcome: Rate of >= Very Good Partial Response (VGPR)
Description: Will be estimated by the number of patients with a VGPR, CR, or Stringent Complete Response (sCR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportions will be calculated.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 40
proportion of participants | 0.74 [0.58 to 0.87] | 0.68 [0.50 to 0.83]

7. Other Pre Specified Outcome: Minor Response Development (MRD)
Description: Will be assessed on bone marrow aspirate in all patients achieving CR. The proportion of patients who achieve MRD negative status will be estimated by the number of patients who are MRD negative divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true MRD negative rate will be calculated.
Time Frame: Up to 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Neurotoxicity
Description: The FACT/GOG neurotoxicity questionnaire will be completed. Patients will be evaluated by overall score for each questionnaire at each time point and changes over time will be calculated. These measures will be correlated with outcome using Fisher's exact test and Kaplan-Meier methods where appropriate.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: All registered patients that were evaluated are included.
Groups:
- Cohort A; Cohort B: MAINTENANCE PHASE: Patients receive ixazomib citrate PO on days 1, 8, and 15 and daratumumab IV over 3-7 hours on day 1. Courses repeat every 28 days for up to 36 months from registration in the absence of disease progression or unacceptable toxicity.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 4/39 | 1/40
Serious Adverse Events (participants affected / at risk) | 10/39 | 8/40
Other Adverse Events (participants affected / at risk) | 39/39 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=39) | Cohort B (N=40)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 2 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=39) | Cohort B (N=40)
Anemia (Blood and lymphatic system disorders) | 4 (9) | 8 (25)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 6 (21)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 24 (212) | 24 (230)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (122) | 21 (167)
Vomiting (Gastrointestinal disorders) | 14 (33) | 13 (53)
Edema limbs (General disorders) | 3 (5) | 1 (4)
Fatigue (General disorders) | 39 (614) | 38 (499)
Pain (General disorders) | 2 (6) | 2 (3)
Infections and infestations - Oth spec (Infections and infestations) | 4 (13) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (3)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (11) | 4 (5)
Upper respiratory infection (Infections and infestations) | 9 (17) | 15 (21)
Urinary tract infection (Infections and infestations) | 8 (10) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (8) | 10 (10)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 8 (60) | 15 (113)
Lymphocyte count decreased (Investigations) | 22 (265) | 27 (282)
Lymphocyte count increased (Investigations) | 4 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 31 (122) | 22 (81)
Platelet count decreased (Investigations) | 23 (149) | 22 (112)
White blood cell decreased (Investigations) | 6 (15) | 15 (50)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 5 (18)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (8) | 3 (11)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (5) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 11 (69) | 3 (60)
Peripheral sensory neuropathy (Nervous system disorders) | 32 (406) | 28 (392)
Presyncope (Nervous system disorders) | 0 (0) | 1 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (2)
Insomnia (Psychiatric disorders) | 7 (15) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (46) | 22 (71)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03012880/Prot_SAP_000.pdf